CLINICAL TRIAL: NCT01456533
Title: Copeptin in the Differential Diagnosis of Dysnatremia in Hospitalized Patients
Acronym: COMED
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Aarau (Other)
Responsible Party: Sponsor
Other Study IDs: COMED Study
Record Dates: First submitted 2011-09-30; First posted 2011-10-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Hyponatremia; Hypernatremia
Keywords: hyponatremia; hypernatremia
MeSH Terms: conditions — Hyponatremia; Hypernatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hospitalized patients: hospitalized patients with hyponatremia

SUMMARY:
Background: Hypo- and hypernatremia are common in hospitalized patients. The differential diagnosis of dysnatremia is challenging.

Osmotically inadequate secretion of antidiuretic hormone (ADH) is the predominant mechanism in most dysnatremic disorders. ADH measurement is cumbersome. It is derived from a larger precursor peptide along with copeptin, which is a more stable peptide directly mirroring the production of ADH.

Objective: To evaluate the additional value of copeptin to improve a currently used algorithm in the differential diagnosis of (A) severe hypoosmolar hypo- and (B) severe hypernatremia.

Design: Prospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* hyponatremia <125 or hypernatremia >155 mmol/L

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with severe hypo or hypernatremia
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of copeptin within hospital stay | participants will be followed for up to 1 year
  diagnostic accuracy will be determined by receiver operated curve (ROC) analysis. The study is powered to detect a difference of copeptin levels between patients with partial central diabetes insipidus (DI) and patients with primary polydipsia.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland; Beat Müller, MD, Principal Investigator — Kantonsspital Aarau, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Mirjam Christ-Crain, Basel, Basel
  - Beat Müller, Aarau, Canton of Aargau

REFERENCES:
- [Derived] Sailer CO, Winzeler B, Nigro N, Bernasconi L, Mueller B, Christ-Crain M. Influence of Outdoor Temperature and Relative Humidity on Incidence and Etiology of Hyponatremia. J Clin Endocrinol Metab. 2019 Apr 1;104(4):1304-1312. doi: 10.1210/jc.2018-01507. PMID 30462243
- [Derived] Nigro N, Winzeler B, Suter-Widmer I, Schuetz P, Arici B, Bally M, Refardt J, Betz M, Gashi G, Urwyler SA, Burget L, Blum CA, Bock A, Huber A, Muller B, Christ-Crain M. Copeptin levels and commonly used laboratory parameters in hospitalised patients with severe hypernatraemia - the "Co-MED study". Crit Care. 2018 Feb 9;22(1):33. doi: 10.1186/s13054-018-1955-7. PMID 29422070